CLINICAL TRIAL: NCT02219373
Title: Gabapentin and Oxcarbazepine for Chronic Neuropathic Pain in Children and Adolescents: A Double-Blind, Randomized Clinical Effectiveness Study.
Brief Title: Gabapentin and Oxcarbazepine for Chronic Neuropathic Pain in Children and Adolescents: A Clinical Effectiveness Study
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Monique Ribeiro, Physician, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P00008001
Record Dates: First submitted 2014-08-08; First posted 2014-08-18 (Estimated); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Pediatric Chronic Neuropathic Pain
MeSH Terms: interventions — Gabapentin; Oxcarbazepine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Gabapentin (Experimental)
  Interventions: Drug: Gabapentin; Other: Placebo
- Oxcarbazepine (Experimental)
  Interventions: Drug: Oxcarbazepine; Other: Placebo
- Placebo (Placebo Comparator): Patients taking placebo will have placebo dose escalated using similar frequency, periods of time, and volumes as those for the active drugs.
  Interventions: Drug: Gabapentin; Drug: Oxcarbazepine; Other: Placebo

INTERVENTIONS:
Drug: Gabapentin — Patients will be randomized to receive either Gabapentin or Oxcarbazepine. The assignment of the medications will be randomized and blinded to both the study investigators and the patient. If patients exhibit >30% pain reduction on receiving the medication evaluated after 4 weeks, then they may continue to receive either the same medication or placebo. If patients exhibit <30% pain reduction, the patient will crossover to the other medication option in the protocol.
  Arms: Gabapentin; Placebo
Drug: Oxcarbazepine — Patients will be randomized to receive either Gabapentin or Oxcarbazepine. The assignment of the medications will be randomized and blinded to both the study investigators and the patient. If patients exhibit >30% pain reduction on receiving the medication evaluated after 4 weeks, then they may continue to receive either the same medication or placebo. If patients exhibit <30% pain reduction, the patient will crossover to the other medication option in the protocol.
  Arms: Oxcarbazepine; Placebo
Other: Placebo — Patients taking placebo will have placebo dose escalated using similar frequency, periods of time, and volumes as those for the active drugs.

SUMMARY:
Given the widespread use of anticonvulsants in the pediatric chronic pain population and the absence of scientific data supporting their use, the investigators propose a randomized, double blind, two group parallel design in which a broad group of children and adolescents with chronic neuropathic pain would be randomized to receive either Gabapentin or Oxcarbazepine.

The Primary Aim of the Study is to assess the frequencies of successful treatment of pediatric patients with neuropathic pain treated with either Gabapentin or Oxcarbazepine.

The Primary Hypotheses are as follows:

Hypothesis I: Both Gabapentin and Oxcarbazepine will result in significant reduction in pain scores when compared to each patient's baseline.

Hypothesis II: Patients who continue on active drug (Gabapentin or Oxcarbazepine) during the second phase of the trial will report greater pain reduction relative to baseline than patients who are randomized onto placebo at this randomization point.

Secondary Aims of the Study are to compare groups treated initially with Gabapentin or Oxcarbazepine with regard to reduction in pain scores (both at rest and with evoked maneuvers), functional disability scores, tolerability, and measures of mood and cognitive functioning.

Secondary Hypotheses are that Gabapentin and Oxcarbazepine differ in their effects on:

1. Pain scores at rest and with evoked maneuvers
2. Functional disability scores
3. Tolerability (frequencies of side-effects)
4. Depression and anxiety scales
5. Neuropsychological measures of cognitive processing speed, working memory, and attention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 8 and 18 at the time of the study with history of chronic (lasting ≥ 4 weeks) neuropathic pain that includes a known injury to a peripheral nerve and/or a pattern of pain responses that includes allodynia, burning, paresthesias or dysesthesias will be included in this study, provided that informed consent has been given by parents.
2. Patient's whose pain rates between moderate to severe at the time of inclusion (ranging from 4-10 in a numeric pain rating scale)
3. Eligible diagnoses include Complex Regional Pain Syndrome, Fibromyalgia, Lumbar Radiculopathy, Spinal Cord Injury, Erythromelalgia, Small Fiber Neuropathies, Traumatic or Post-surgical Peripheral Nerve or Plexus Injuries, and Extremity Pain with severe pain to light touch (allodynia).
4. Child has age-appropriate spoken and written knowledge of English.
5. Parent may be able to utilize an interpreter if need be.

Exclusion Criteria:

1. Unstable psychiatric illness (suicidal ideation, disorganized behavior)
2. Uncontrolled Seizure disorder
3. Chronic Headaches only
4. Abdominal Pain only
5. Prior experience with anticonvulsants for pain treatment.
6. Patients with Syndrome of Inappropriate Secretion of Antidiuretic Hormone

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
As a primary outcome, success will be defined by clinically and statistically significant within subject reductions in pain scores | 0 (baseline), 2, 4, 6, 8 weeks (post-assignment of intervention)
  1. 2 point reduction in average daily pain scores
  2. 30% reduction relative to baseline
  3. Global overall impression of strong benefit.

SECONDARY OUTCOMES:
Pain Scores at rest and evoked maneuvers | 0 (baseline) and 4 and 8 weeks (post assignment of intervention)
  The investigators will assess pain scores at rest and with evoked maneuvers through exam and quantitative sensory test.
Frequency of side effects- Tolerability | 1, 2, 4, 6, 8 weeks (post assignment of intervention)
  * Common side effects include headaches and feeling sleepier in the morning and having less energy. Side effects that can occur, but are not common, include gastrointestinal side effects (upset stomach or throwing up, diarrhea or constipation, and weight gain), feeling lightheaded, having blurred eyesight, shakiness or changes in balance.
  * Very rarely, patients taking these medicines may experience memory problems, sadness, nervousness, and Serious Adverse Events (SAEs).
  Routine laboratory testing will be conducted as part of the safety profile assessment.
Functional Disability Scores | 0 (baseline), 4, and 8 weeks (post-assignment of intervention)
Frequency of Side effects- Depression and Anxiety | Baseline, Week 4 and 8 (post assignment of the intervention)
  As both study medicines may be associated with mood changes and as pain itself sometimes is co-morbid with anxiety and depression, the investigators will perform self-report measures of anxiety and depression (Children's Depressive Inventory and The Revised Children's Manifest Anxiety Scale) pre and post-assigment of the intervention.
Frequency of Side Effects- Neuropsychological Measures | Baseline, weeks 4 and 8 (post-assignment of the intervention).
  Both study medicines may be associated with the emergence of cognitive side effects to include difficulties with concentration and cognitive slowing. The investigators will assess for cognitive processing speed, working memory and attention difficulties during the course of treatment using the NIH toobox Cognitive Battery.

CONTACTS AND LOCATIONS:
Overall Officials: Monique Ribeiro, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States